CLINICAL TRIAL: NCT00544336
Title: Assessment of Family Quality of Life Among Families With a Member Who is a Cancer Patient
Brief Title: Family Quality of Life Among Families With a Member Who is a Cancer Patient
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine; Director, Cancer Supportive Care Program; Director, Head and Neck Research Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC SUPP 0737; VU-VICC-SUPP-0737; VU-VICC-IRB-IRB-070598
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer; Colorectal Cancer; Head and Neck Cancer; Lung Cancer; Prostate Cancer; Solid Tumor
Keywords: unspecified adult solid tumor, protocol specific; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent non-small cell lung cancer; recurrent small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage I adenoid cystic carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; stage I basal cell carcinoma of the lip; stage II basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; high-grade salivary gland mucoepidermoid carcinoma; low-grade salivary gland mucoepidermoid carcinoma; recurrent salivary gland cancer; salivary gland acinic cell tumor; salivary gland adenocarcinoma; salivary gland adenoid cystic carcinoma; salivary gland anaplastic carcinoma; salivary gland malignant mixed cell type tumor; salivary gland poorly differentiated carcinoma; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Colonic Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Supportive
  Interventions: Other: questionnaire administration; Other: survey administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: questionnaire administration — no intervention
Other: survey administration — no intervention
Procedure: quality-of-life assessment — no intervention

SUMMARY:
RATIONALE: Developing a questionnaire that can be used to assess the quality of life among people who have a family member with cancer may help the study of cancer in the future.

PURPOSE: This clinical trial is studying quality of life among families with a member who is a cancer patient.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop and conduct preliminary validation of a Family Quality of Life Questionnaire for use with families with an adult cancer patient, with the measure appropriate for use for both research and clinical assessment purposes.
* Generate an initial item pool for the measure (step 1).
* Reduce the item pool based on a content validity assessment (step 2).
* Assess the psychometric properties and dimensionality of the measure (step 3).

OUTLINE:

* Step 1 (item generation): Items are generated through a literature review and a semi-structured interview with patients and their families. The purposes of the interview are to determine whether the five domains identified in the literature review (family interaction, family roles, family communication, family emotional support, overall family quality of life [FQOL]) are central areas of FQOL, and to determine if there are other important FQOL domains affected by cancer and its treatment. Patients and their family members are interviewed individually over 45-60 minutes. The initial item pool is generated based on the literature review and interviews.
* Step 2 (item review and reduction): The initial item pool is examined and reduced based on its content validity. Ten health care providers with a minimum of five years experience working with cancer patients rate the content validity of the proposed questionnaire. Experts receive a packet of questionnaires, including the objective of the study, the proposed questionnaire as developed in step 1, and the proposed questionnaire with its format modified for the examination of content validity. The content validity version uses a 4-point Likert format to assess each item's relevance, sufficiency (i.e., the extent to which it fully covers its intended domain) and clarity in relation to the construct (FQOL domain) that it is supposed to assess. Experts are asked to rate the overall format of the questionnaire in regards to ease of use and appropriateness, and for open-ended comments or suggestions. Items are modified or dropped based on the experts' review.
* Step 3 (final item selection and psychometric evaluation): Patients and family members complete the FQOL questionnaire developed in previous steps and other questionnaires with proven reliability and validity at baseline. Other questionnaires include the SF-36 (general QOL survey that is used widely in general population samples and patients, including cancer patients), the FACT-G for patients (instrument used to assess health-related QOL in cancer patients), with the version of the FACT-G modified by Northouse for the family member, the Family Interaction and Emotional Well-Being subscales (to examine family interaction and family emotional support of cancer families) of the Beach Center Family Quality of Life Scale (FQOL measure for families with a disabled child), the Balanced Cohesion subscale (to examine family interaction of cancer families) of the FACES IV (that assesses balanced and unbalanced family cohesion and family flexibility in general population), and the Family Communication Scale (a general survey used to assess family communication in the general population). Patients and family members complete the FQOL again 2 weeks after the initial assessment.

PROJECTED ACCRUAL: Approximately 210 cancer patients and 210 family members will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with any local, advanced, or metastatic cancer that has required more than a simple surgical procedure

  * Ten families with an adult patient with breast, prostate, lung, colon, or head and neck cancer are interviewed for step 1 portion of the study
* An available adult family member willing to participate in the study

  * The term family is defined broadly to include adults over 21 years of age, considered by the cancer patient as a family member, who provides care or support and/or shares the cancer experience with the patient
  * Family members do not need to be biologically related to the patient or related through marriage, and may or may not live in the same house with the patient

Exclusion Criteria:

* Able to read, write, and speak English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Family members of a patient with cancer
Sampling Method: Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Preliminary validation of a family quality of life questionnaire | Off study date
Generation of an initial item pool (step 1) | Off study date
Reduction of the item pool based on content validity assessment (step 2) | Off study date
Psychometric properties and dimensionality of the measure (step 3) | Off study date

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee